CLINICAL TRIAL: NCT02530151
Title: Prospective Assessment of Intraoperative Intra-articular Morphine and Clonidine Injection in Hip Arthroscopy on Postoperative Pain Management
Brief Title: Intra-articular Morphine and Clonidine Injections for Pain Management in Hip Arthroscopy
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Northwestern University (Other)
Responsible Party: Principal Investigator, Michael Terry, Associate Professor in Orthopaedic Surgery, Northwestern University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Supportive Care
Other Study IDs: STU00201218
Record Dates: First submitted 2015-08-18; First posted 2015-08-20 (Estimated); Results first posted 2019-05-20 (Actual); Last update posted 2019-09-23 (Actual); Status verified 2019-09

CONDITIONS: Femoracetabular Impingement; Pain, Postoperative
Keywords: Hip arthroscopy; Intra-articular injection; Morphine; Clonidine
MeSH Terms: conditions — Femoracetabular Impingement; Pain, Postoperative | interventions — Morphine; Clonidine; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Morphine with Clonidine (Experimental): 11 mL intra-articular injection of 10 mg morphine and 100 mcg clonidine in .9% NaCl solution at conclusion of hip arthroscopy procedure
  Interventions: Drug: Morphine with clonidine
- Normal Saline (Placebo Comparator): 11 mL intra-articular injection of .9% NaCl solution at conclusion of hip arthroscopy procedure
  Interventions: Other: Normal saline

INTERVENTIONS:
Drug: Morphine with clonidine — see arm description
  Arms: Morphine with Clonidine
Other: Normal saline — see arm description
  Arms: Normal Saline

SUMMARY:
The purpose of this study is to determine whether intraoperative (during surgery) morphine and clonidine hip injections are effective in postoperative pain management for patients undergoing hip arthroscopy.

DETAILED DESCRIPTION:
Background:

Over the last few decades, the use and safety of arthroscopic hip surgery has considerably improved though the evolution and development of arthroscopic imaging and instrumentation (Lynch et al., 2013). There is still a considerable amount of room for growth and research in comparison to arthroscopic knee and shoulder surgery, which have been around much longer. One area which needs attention is postoperative pain management for patients undergoing hip arthroscopy. The benefits to controlling postoperative pain range from improved patient comfort and decreased time of recovery to decreased narcotic medication usage and reduced cost of care (Ramsay 2000).

Many studies on the use of morphine injections into the joint after arthroscopic knee surgery have demonstrated effectiveness in reducing both patient reported pain and narcotic medication usage after surgery (Stein et al., 1991; Yari et al., 2013; Zeng et al., 2014). Furthermore, studies have shown that joint injections of clonidine improve the pain relieving effect of morphine when the two are used in combination (Joshi et al., 2000). While there is considerable evidence supporting the use of joint injections of morphine for knee surgery, very little has been cited for such use in hip arthroscopy (Lavelle et al., 2007). The purpose of our study is to better assess the effectiveness of morphine and clonidine joint injections in reducing patient reported pain and narcotic medication usage after hip arthroscopy.

Protocol:

Participants in this study will be part of a trial for the use of a morphine and clonidine joint injection during hip surgery. Participants will be randomly selected to either receive a standard dose of morphine and clonidine or normal saline solution through a joint injection. The normal saline will have no active drug ingredients. In either case the injection will occur at the conclusion of surgery. The joint injection is the only change to the medical care that will occur for patients who decide to participate in this study. Pain levels will be monitored and treated after surgery, and all pain management after surgery will follow the normal standard of care. Additionally, participants will be asked to fill out a brief questionnaire before and after surgery. All patients will be sent home with a short diary that will allow them to record their medication usage, pain scores, and potential side effects in the week following surgery. The diary with this information will be returned when the patients come back for their standard-of-care two week follow-up appointment.

No additional visits or appointments beyond what the procedure already entails are needed to participate in this study.

The treatment (morphine/clonidine or normal saline injection) will be chosen by chance, like flipping a coin. Neither the participant nor the study doctor will choose which treatment the patient gets. There will be an equal chance of being given either treatment. Neither the participant nor the study doctor will know which treatment is assigned.

Morphine and clonidine are FDA-approved drugs being used in a non-approved context (hip injection). All standard of care procedures will take place to ensure patient safety during and after surgery, while the patients are in the outpatient surgical center. All adverse events will be properly documented and reported to the IRB.

Data Management:

Data points include age, sex, height, weight, tobacco use, VAS pain scores, discharge times, duration of surgery, discharge criteria score, medication use, and scores from the QoR-15 survey. All information that includes personally identifying information, such as name or medical record number, is not entered into the database with the medical information. Identifying information is only entered into a separate database that links the patient to an arbitrary study number.

Statistical analysis of the data will include a Student's T-Test, non-parametric Mann Whitney test, and chi-square test. If there is substantial data missing for a subject, which would be otherwise essential for analysis, the subject's information for that particular analysis will be excluded. To the best extent possible, data that can be interpolated will be utilized.

ELIGIBILITY:
Inclusion Criteria:

* Any patient undergoing a hip arthroscopy procedure for femoracetabular impingement by the senior surgeon (M.T.)

Exclusion Criteria:

* Morphine contraindication
* Clonidine contraindication
* Pregnant women
* Prisoners
* Adults unable to consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2015-11; Primary Completion 2017-05 (Actual); Study Completion 2017-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael Terry, MD, Principal Investigator — Northwestern University
Locations (1):
- Joshua Barett, Chicago, Illinois, United States

REFERENCES:
- [Background] Lynch TS, Terry MA, Bedi A, Kelly BT. Hip arthroscopic surgery: patient evaluation, current indications, and outcomes. Am J Sports Med. 2013 May;41(5):1174-89. doi: 10.1177/0363546513476281. Epub 2013 Feb 28. PMID 23449836
- [Background] Ramsay MA. Acute postoperative pain management. Proc (Bayl Univ Med Cent). 2000 Jul;13(3):244-7. doi: 10.1080/08998280.2000.11927683. No abstract available. PMID 16389390
- [Background] Stein C, Comisel K, Haimerl E, Yassouridis A, Lehrberger K, Herz A, Peter K. Analgesic effect of intraarticular morphine after arthroscopic knee surgery. N Engl J Med. 1991 Oct 17;325(16):1123-6. doi: 10.1056/NEJM199110173251602. PMID 1653901
- [Background] Yari M, Saeb M, Golfam P, Makhloogh Z. Analgesic efficacy of intra-articular morphine after arthroscopic knee surgery in sport injury patients. J Inj Violence Res. 2013 Jul;5(2):84-8. doi: 10.5249/jivr.v5i2.303. Epub 2013 Jul 1. PMID 23281420
- [Background] Zeng C, Gao SG, Cheng L, Luo W, Li YS, Tu M, Tian J, Xu M, Zhang FJ, Jiang W, Wei LC, Lei GH. Single-dose intra-articular morphine after arthroscopic knee surgery: a meta-analysis of randomized placebo-controlled studies. Arthroscopy. 2013 Aug;29(8):1450-8.e2. doi: 10.1016/j.arthro.2013.04.005. Epub 2013 Jun 12. PMID 23768848
- [Background] Joshi W, Reuben SS, Kilaru PR, Sklar J, Maciolek H. Postoperative analgesia for outpatient arthroscopic knee surgery with intraarticular clonidine and/or morphine. Anesth Analg. 2000 May;90(5):1102-6. doi: 10.1097/00000539-200005000-00018. PMID 10781460
- [Background] Lavelle W, Lavelle ED, Lavelle L. Intra-articular injections. Anesthesiol Clin. 2007 Dec;25(4):853-62, viii. doi: 10.1016/j.anclin.2007.07.002. PMID 18054149

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Morphine With Clonidine | Normal Saline
Started | 37 | 33
Completed | 16 | 17
Not Completed | 21 | 16

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Morphine With Clonidine | Normal Saline | Total
Number analyzed (Participants) | 37 | 33 | 70
Age, Continuous [Mean (Standard Deviation); unit: years] | 40.7 (12.9) | 36.7 (11.8) | 38.8 (12.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 25 | 19 | 44
  Male | 12 | 14 | 26
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 37 | 33 | 70
Smoking Status [Count of Participants; unit: Participants]
  No | 35 | 30 | 65
  Yes | 2 | 3 | 5
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kg/m^2] | 25.8 (3.5) | 25.5 (3.8) | 25.6 (3.6)
Surgical duration [Mean (Standard Deviation); unit: minutes] | 43.9 (13.7) | 42.4 (9.5) | 43.2 (11.7)
Concomitant Procedures [Count of Participants; unit: Participants]
  Iliopsoas lengthening | 5 | 11 | 16
  IT band windowing/trochanteric bursectomy | 11 | 6 | 17
  Loose body removal | 0 | 1 | 1
Time to recovery [Mean (Standard Deviation); unit: minutes] | 172 (40.5) | 172 (42) | 172 (41.2)

OUTCOME MEASURES:

1. Primary Outcome: Opioid Consumption in the Acute Postoperative Period
Description: The total usage of opioid medication (mEq) for pain relief in the intraoperative period and again through the postoperative recovery period from arrival in the PACU through 7 days post op
Time Frame: Recorded intraoperatively, during PACU stay, 6 hours post discharge, 18 hours post discharge, 24 hours post discharge, 48 hours post discharge, and at 7 days post discharge
Population: Patients that failed to complete the necessary follow up for all time points following discharge (6 hrs/18 hrs/24 hrs/48 hrs) were excluded from final analysis for the respective time points
Measure: Mean (95% Confidence Interval); unit: milligram morphine equivalents (mEq)
Arm/Group | Morphine With Clonidine | Normal Saline
Number analyzed (Participants) | 37 | 33
milligram morphine equivalents (mEq)
  Intraoperative | 57.3 [50.6 to 63.9] | 56.0 [47.6 to 64.4]
  PACU | 37.0 [28.8 to 45.3] | 40.1 [31.8 to 48.4]
  6 hours Post Discharge: number analyzed (Participants) | 17 | 16
  6 hours Post Discharge | 5.5 [3.7 to 7.3] | 5.3 [3.0 to 7.6]
  18 hours Post Discharge: number analyzed (Participants) | 17 | 16
  18 hours Post Discharge | 14.5 [10.6 to 18.4] | 13.8 [8.7 to 18.9]
  24 hours Post Discharge: number analyzed (Participants) | 17 | 16
  24 hours Post Discharge | 19.5 [13.9 to 25.1] | 20.0 [12.1 to 27.8]
  48 hours Post Discharge: number analyzed (Participants) | 17 | 16
  48 hours Post Discharge | 27.7 [19.5 to 35.9] | 35.6 [18.3 to 52.9]
  7 days Post Discharge: number analyzed (Participants) | 17 | 16
  7 days Post Discharge | 50.7 [29.6 to 71.7] | 73.8 [31.6 to 115.9]

2. Secondary Outcome: Visual Analog Scale (VAS) Pain Scores
Description: Patients will rate their pain (0-10) on the Visual Analog Scale with higher scores for the VAS indicated elevated pain intensity reported by the patient for the indicated time point
Time Frame: Immediately preoperative (5-10 minutes before surgery), immediately postoperative (5-10 minutes after surgery), 1 hr post operatively
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Morphine With Clonidine | Normal Saline
Number analyzed (Participants) | 37 | 33
score on a scale
  Preoperative VAS Pain Score | 2 [1 to 3] | 2 [1 to 3]
  Immediate Post Op VAS Pain Score | 3 [2 to 4] | 4 [3 to 5]
  1 hr. Post Op VAS Pain Score | 4 [3 to 5] | 5 [4 to 5]

3. Secondary Outcome: Quality of Recovery (QoR-15) Scores for Patient Reported Recovery Following Surgery
Description: The Quality of Recovery questionnaire (QoR-15) is a 15 question patient reported outcome measure used to evaluate the quality of recovery following surgical anesthesia concerning pain, physical function, and psychological factors; reported as a summative score with each question graded between 0-10 (Range:0-150) with higher scores indicating improved physical/psychological recovery or infrequent symptoms
Time Frame: Preoperative to 24 hrs. post operatively
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Morphine With Clonidine | Normal Saline
Number analyzed (Participants) | 37 | 33
score on a scale
  Preoperative QoR-15 Score | 123 [108 to 138] | 131 [125 to 137]
  Change in QoR-15 Score at 24 hrs. Post Op | -22 [-35 to -9] | -20 [-29 to -10]

ADVERSE EVENTS:
Description: Adverse events were not monitored or assessed for any study participants due to the nature of the hip arthroscopy procedure and the study procedures at large
Arm/Group | Morphine With Clonidine | Normal Saline
All-Cause Mortality (participants affected / at risk) | 0/0 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2015-10-23): https://cdn.clinicaltrials.gov/large-docs/51/NCT02530151/Prot_SAP_000.pdf
  • Informed Consent Form (2015-10-30): https://cdn.clinicaltrials.gov/large-docs/51/NCT02530151/ICF_001.pdf